CLINICAL TRIAL: NCT02829333
Title: Effect of Anesthetic Technique on Serum Vascular Endothelial Growth Factor C and Prostaglandin E2 in Women Undergoing Surgery for Uterine Leiomyomas
Brief Title: The Effect of Anesthetic Technique on VEGF-C and PGE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Zhangyonghai001
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2016-07

CONDITIONS: Uterine Leiomyomas
Keywords: analgesia; anesthesia; leiomyomas; tumor; vascular endothelial growth factor; anesthesia technique on tumor
MeSH Terms: conditions — Myofibroma; Agnosia; Leiomyoma; Neoplasms | interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group GA (Other): 22 patients receive general anesthesia and patient controlled intravenous analgesia
  Interventions: Other: general anesthesia and patient controlled intravenous analgesia
- Group SA (Other): 22 patients receive spinal anesthesia and continuous postoperative epidural analgesia
  Interventions: Other: spinal anesthesia and continuous postoperative epidural analgesia

INTERVENTIONS:
Other: general anesthesia and patient controlled intravenous analgesia — Patients receive general anesthesia intraoperative period and continuous intravenous analgesia postoperation
  Arms: Group GA
Other: spinal anesthesia and continuous postoperative epidural analgesia — Patients receive spinal anesthesia intraoperative period and continuous epidural analgesia postoperation
  Arms: Group SA

SUMMARY:
The purpose of this study is to verify the effect of anesthetic technique on the change of postoperative serum vascular endothelial growth factor C and prostaglandin E2, and to explore the potential impact of the anesthetic technique on leiomyomas recurrence and growth after the surgery of abdominal myomectomy.

DETAILED DESCRIPTION:
Uterine leiomyomas is the most common benign tumor of uterus, the most common tumor in women as well. Like many other forms of tumor, it requires an independent blood supply to enlarge. This process, angiogenesis, is mediated by vascular endothelial growth factor C (VEGF-C) and prostaglandin E2 (PGE2). Several studies have confirmed that VEGF-C has a high level in patients with uterine leiomyomas, which has also been demonstrated that it was related to occurrence and growth of uterine leiomyomas because it's capable of promoting angiogenesis, mitogenic, and vascular permeability-enhancing activities. Also, some researchers suggested that suppression of prostaglandin synthesis (including PGE2) via cyclooxygenase type-2 (COX-2) enzyme inhibition may reduce the incidence of some tumor. The aim of this study is to verify the effect of anesthetic technique on the change of postoperative serum VEGF-C and PGE2, and to explore the potential impact of the anesthetic technique on leiomyomas recurrence and growth after the surgery of abdominal myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* The patients with leiomyomas requiring abdominal myomectomy, aged 18-65 year and American Society of Anesthesiologists (ASA) physical status I or II.

Exclusion Criteria:

* The patients who had a history of surgery within the preceding two weeks, a history of blood transfusion and a history of coronary artery disease, any contraindication to spinal anesthesia or opioid analgesia.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change of vascular endothelial growth factor C before anesthesia and at 48 hours after surgery | Before anesthesia and at 48 hours after surgery
  Blood samples were sampled before anesthesia and at 48h after surgery for the serum VEGF-C，which were analyzed by using enzyme linked immunosorbent assay (ELISA).
Change of prostaglandin E2 before anesthesia and at 48 hours after surgery | Before anesthesia and at 48 hours after surgery
  Blood samples were sampled before anesthesia and at 48h after surgery for the serum PGE2，which were analyzed by using enzyme linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Visual analog scale (VAS) pain scores | at 2h, 4h, 8h, 12h, 24h and 48h after surgery
  Visual analog scale (VAS) pain scores were used to evaluate postoperative pain at 2h, 4h, 8h, 12h, 24h and 48h after surgery by the anesthetist

IPD SHARING:
Plan to Share IPD: No